CLINICAL TRIAL: NCT01060748
Title: Development of a Polyvalent Vaccine Against Enterotoxigenic Escherichia Coli (ETEC)Protective Efficacy of the Deletion-Attenuated, Multi-valent ACE527 Against Challenge With a Prototype Strain of Enterotoxigenic E.Coli Expressing LT and ST Enterotoxins and CFA/I (Strain H10407) in Human Challenge Model.
Brief Title: Safety and Efficacy Study of a Vaccine Against Enterotoxigenic Escherichia Coli (ETEC) to Prevent Moderate to Severe Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TD Vaccines A/S (Industry)
Collaborators: Pierrel Research USA, Inc. (Industry); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Ingelise Saunders/CEO, TD Vaccines A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACE527-102
Record Dates: First submitted 2010-01-28; First posted 2010-02-02 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Diarrhea
Keywords: Vaccination; Challenge; Diarrhea; ETEC illness; Travelers diarrhea; ETEC; Enterotoxigenic E.coli
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACE527 (Experimental): First cohort: ACE527 vaccine doses of 9 x 10E10 cfu on study day 0 and 21 on an outpatient basis.
  Second cohort: ACE527 vaccine dose of 9 x 10E10 cfu on study day 0 and 21 on an outpatient basis.
  Interventions: Biological: ACE527
- Placebo vaccine (Placebo Comparator): First cohort: Placebo vaccine on study day 0 and 21 on an outpatient basis.
  Second cohort: Placebo vaccine on study day 0 and 21 on an outpatient basis.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ACE527 — ACE527 comprises a mixture of three live, attenuated ETEC strains; ACAM2025 (CFA/I+ and LTB+), ACAM2022 (CS5+, CS6+ and LTB+), and ACAM2027 (CS1+, CS2+, CS3+ and LTB+). The vaccine is administered orally as a two-dose regimen, at 9x1010 cfu, on Days 0 and 21, in 200 ml CeraVacx buffer. The required volume of each vaccine strain, supplied as a frozen suspension, is mixed into the buffer solution prior to dosing.
  Arms: ACE527
Biological: Placebo — Placebo
  Arms: Placebo vaccine

SUMMARY:
This is a research study about an experimental (investigational) vaccine called ACE527. ACE527 is a vaccine that is being made to prevent disease from a germ called enterotoxigenic Escherichia coli (ETEC). This germ causes diarrhea, largely in children living in developing countries and in travelers to those countries. One purpose of this study is to see if the vaccine is safe and develops an immune response. Another purpose is to see if it prevents people from getting sick when exposed to the ETEC germ. This ETEC germ is also experimental (investigational).

DETAILED DESCRIPTION:
This is a single-center, double-blind, placebo-controlled, Phase II vaccination and challenge study designed to assess the protective efficacy of the ACE 527 vaccine, as well as collect expanded safety and immunogenicity data. The study will be carried out in two phases. In the initial vaccination phase, up to 72 subjects will be randomized 1:1 to receive either ACE527 or placebo on an outpatient basis. Vaccine and placebo preparations will be given orally. Following vaccination, subjects will be followed as out-patients for safety using diary card surveillance, for vaccine shedding by qualitative stool culture (i.e. presence or absence) and for the development of local and systemic antibody responses to the ACE527 vaccine strains. In the subsequent inpatient challenge phase, up to 56 vaccinated subjects will be admitted as inpatients and challenged with the ETEC strain, H10407. The challenge dose will be administered orally.After challenge, subjects will be monitored for diarrhea and other signs/symptoms of enteric illness by daily medical checks, vital sign determinations, grading and weighing of all stools. Monitoring for fecal shedding of the challenge ETEC strain H10407 will occur daily, after challenge, while in-patient. Local and systemic antibody responses to the challenge ETEC strain H10407 will also be assessed. All subjects will be treated with Abx.

ELIGIBILITY:
Inclusion criteria:

* Male or female age ≥18 and ≤ 50 years.
* General good health, without clinically significant medical history, physical examination findings or clinical laboratory abnormalities per clinical judgment of PI.
* Negative serum pregnancy test before first (visit V0) and before challenge (visit C0) for female subjects of childbearing potential. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable. Female subjects unable to bear children must have this documented (e.g. tubal ligation or hysterectomy) or must have negative pregnancy tests.
* Willingness to participate in the study after all aspects of the protocol have been explained and written informed consent obtained.
* Completion of a training session and demonstrated comprehension of the protocol procedures, knowledge of ETEC-associated illness, and by passing a written examination.
* Availability for the study duration, including all planned follow-up visits.

Exclusion criteria:

* Presence of a significant medical or psychiatric condition which in the opinion of the investigator precludes participation in the study. Some medical conditions which are adequately treated and stable would not preclude entry into the study. These conditions might include stable asthma controlled with inhalers or mild hypertension stably controlled with a single agent.
* Significant abnormalities in screening hematology, serum chemistry or urinalysis as determined by PI or PI in consultation with the MM and sponsor.
* Presence in the serum of HIV antibody, HBsAg, or HCV antibody.
* Evidence of IgA deficiency (serum IgA < 7 mg/dl or limit of detection of assay).
* Evidence of current excessive alcohol consumption or drug dependence.
* Evidence of impaired immune function.
* BMI <19, >34
* Recent vaccination or receipt of an investigational product (within 30 days before vaccination).
* Intention to donate blood or blood products for one month following the completion of study participation (note: The Red Cross will not allow blood donations for 1 year following participation in an investigational research study).
* Any other criteria which, in the investigator's opinion, would compromise the ability of the subject to participate in the study, the safety of the study, or the results of the study
* Working as a food handler, in child-care or as a healthcare worker with direct patient contact.
* Have household contacts who are <2 years old or >80 years old or infirm or immunocompromised (for reasons including corticosteroid therapy, HIV infection, cancer chemotherapy, or other chronic debilitating disease).
* Abnormal stool pattern (fewer than 3 per week or more than 3 per day).
* Regular use of laxatives, antacids, or other agents to lower stomach acidity.
* Use of any medication known to affect the immune function (e.g., corticosteroids and others) within 30 days preceding the first vaccination or planned use during the active study period.
* Known allergy to two of the following antibiotics: quinolones, trimethoprim-sulfamethoxazole, and penicillin.
* Symptoms consistent with Traveler's Diarrhea concurrent with travel to countries where ETEC infection is endemic (most of the developing world) within two years prior to dosing, OR planned travel to endemic countries during the length of the study.
* Vaccination for or ingestion of ETEC, cholera, or LT toxin within 3 years prior to dosing.
* Use of antibiotics during the 7 days before dosing or proton pump inhibitors, H2 blockers or antacids within 48 hours prior to dosing.
* History of diarrhea in the 7 days prior to vaccination (outpatient diarrhea is defined as ≥ 3 unformed loose stools in 24 hours).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Severe diarrhea: ≥6 grade 3-5 stools in 24 hrs, or >800g of grade 3-5 stools in 24 hrs and moderate diarrhea: 4-5 grade 3-5 stools in 24 hrs or 401-800g of grade 3-5 stools in 24 hrs | Study Day 49 to 57

SECONDARY OUTCOMES:
Number of subjects with severe diarrhea (if any) | Study Day 49 to 57
Number of subjects with diarrhea of any severity | Study Day 49 to 57
Mean total weight of grade 3-5 stools passed per subject | Study Day 49 to 57
Mean number of grade 3-5 stools per subject | Study day 49 to 57
Number of subjects with nausea, vomiting, anorexia, or abdominal pain/cramps rated as moderate to severe. | Study Day 0 to 77
Number of subjects who indicate they would have reduced their daily activity if they had been vacationing or traveling for business because of their ETEC illness. | Last visit
Mean time to onset of diarrhea. | Study Day 49 to 57
Number of subjects with moderate to severe ETEC illness | Study Day 49 to 57
Number of colony forming unite (cfu) of the challenge strain per gram of stool | Study day 49 to 57
Number of subjects requiring early antibiotic treatment | Study Day 49 to 57
Number of subjects requiring IV fluids | Study Day 49 to 57
Systemic immune responses to the constituent strains of the vaccine | Selected Time Points
Mucosal immune responses to the constituent strains of the vaccine | Selected Time Points
The intestinal colonization by the three individual vaccine strains and challenge strain post-vaccination | Selected Time Points

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Harro, MD, Principal Investigator — CIR, Johns Hopkins School of Public Health
Locations (1):
- Center for Immunization Research (CIR), Baltimore, Maryland, United States